CLINICAL TRIAL: NCT03128216
Title: Comparison of Local Anesthetic Infiltration, Trasversalis Fascia Block or Spinal Anesthesia for Inguinal Hernia Repair
Brief Title: Local Anesthetic Infiltration VS Trasversalis Fascia Block VS Spinal Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istituti Ospitalieri di Cremona (Other)
Responsible Party: Principal Investigator, Erika Basso Ricci, Principal Investigator, Istituti Ospitalieri di Cremona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANECR_02_17
Record Dates: First submitted 2017-04-12; First posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Anesthesia, Spinal; Ropivacaine; Bupivacaine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blind Local Anesthetic Infiltration (Active Comparator)
  Interventions: Procedure: Blind Local Anesthetic infiltration; Drug: Ropivacaine
- Transversals Fascia Block (Active Comparator)
  Interventions: Procedure: Transversals Fascia Block; Drug: Ropivacaine
- Spinal Anesthesia (Active Comparator)
  Interventions: Procedure: Spinal Anesthesia; Drug: Bupivacaine

INTERVENTIONS:
Procedure: Blind Local Anesthetic infiltration — Patients of this group received blind local anesthetic infiltration on surgical site. Local anesthetic infiltration are performed by surgeon.
  Arms: Blind Local Anesthetic Infiltration
Procedure: Transversals Fascia Block — Patients of this group received ultrasound guided omolateral Transversals Fascia Block.
  Arms: Transversals Fascia Block
Procedure: Spinal Anesthesia — Patients of this group received Spinal Anesthesia
  Arms: Spinal Anesthesia
Drug: Ropivacaine — Local anesthetic used for local infiltration and Transversals fascia block
  Arms: Blind Local Anesthetic Infiltration; Transversals Fascia Block
Drug: Bupivacaine — Local anesthetic used for Spinal Anesthesia
  Arms: Spinal Anesthesia

SUMMARY:
Propose to comparison effectiveness of blind local anesthetic infiltration with ultrasound guided Transversals Fascia Block and Spinal Anesthesia in patients undergoing to inguinal hernia repair surgery. The effectiveness is defined as pain control during intraoperative and time need to reach hospital discharge criteria in the post-operative period.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years;
* ASA score I - II - III;
* patients undergoing elective inguinal hernia repair;
* signed informed consent;

Exclusion Criteria:

* chronic therapy with opioids/ antidepressants;
* urgent/emergent surgery;
* postoperative transfer to the intensive care unit;
* known allergy to any drug medication;
* local skin infection;
* epilepsy;
* alcohol or drug abuse;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Hospital discharge | First 6 post-operative hours
  Time need to reach hospital discharge criteria in post-operative period

SECONDARY OUTCOMES:
Intraoperative Pain Control | Intraoperative period
  Need of addiction local anesthetic or endovascular anesthetic to performed surgery
Post-operative Pain | Post-operative period for 6 hours, every 30 min
  NRS score in post-operative period
Side effects | intra-operative and post-operative period (6 hours)
  Incidence of side effects
Chronic Pain | at 1 week and 3 months in post-operative period
  Incidence of chronic post-operative pain

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Cremona, Creom, Cremona, Italy

IPD SHARING:
Plan to Share IPD: No